CLINICAL TRIAL: NCT03156894
Title: Heart Transplant and Primary Transplant Dysfunction: a Retrospective Analysis of the Strasbourg Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 6733
Record Dates: First submitted 2017-01-04; First posted 2017-05-17 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2017-05

CONDITIONS: Primary Graft Dysfunction
Keywords: Graft Dysfunction; Primary Graft Dysfunction; heart transplant; heart failure; Hemodynamic parameters; Incidence of PDG
MeSH Terms: conditions — Primary Graft Dysfunction; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Among the complications of heart transplant, primary dysfunction of the graft (PDG) is the most feared with a net impact on early morbidity and mortality. The all-cause mortality rate at the international level is 10% at 30 days and 34% at one year. Mortality at 30 days is secondary in 66% of cases with DPG or multi-organ failure.

The treatment of choice for the more severe PDG remains ECMO-type circulatory mechanical assistance or ventricular assistance. According to several studies, this could reduce early mortality. Early placement and short-term (<30 days) of support appear to improve survival in the first year after transplantation.

The haemodynamic parameters revealing this DPG are not clearly described in the literature.

hypothesis of this research is that:

* DPG risk factors in strasbourg's hospital center are comparable to other European and international centers.
* Simple hemodynamic parameters can be used to detect PDG earlier in order to set up assistance more quickly.

ELIGIBILITY:
Inclusion Criteria:

* All patients who had an isolated heart transplant in the cardiac surgery department of HUS (Hôpitaux Univertsitaires de Strasbourg) between June 2008 and December 2015.

Exclusion Criteria:

* multi-organ transplants, patients with secondary graft dysfunction and those whose postoperative data were not accessible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who had an isolated heart transplant in the cardiac surgery department of HUS (Hôpitaux Univertsitaires de Strasbourg) between June 2008 and December 2015.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
Retrospective comparison of risk factors (incidence for ordinal and average variables for numerical variables) between patients suffering from severe primary dysfunction of the graft and those not suffering from severe primary dysfunction of the graft | 1 month after leaving the operating room

CONTACTS AND LOCATIONS:
Locations (1):
- Service Réanimation chirurgicale cardio-vasculaire - NHC, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No